CLINICAL TRIAL: NCT04135261
Title: A Phase 1 Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of HBM4003 in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerance and Anti-tumor Activity of a Study Drug in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbour BioMed US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4003.1
Record Dates: First submitted 2019-10-15; First posted 2019-10-22 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumors

STUDY DESIGN:
Intervention Model Description: Dose escalation (Part 1) followed by Dose expansion (Part 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose escalation (Experimental): QW - up to 4 (28 day) cycles of treatment (treatment administered 1x weekly) or Q3W - up to 6 (21 day) cycles of treatment (treatment administered 1x q3w)
  Dose for cohorts to be confirmed following consultation and approval by Safety Review Committee.
  Interventions: Drug: HBM4003
- Part 2: Dose expansion (Experimental): Treatment administered at Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) established in Part 1, in specific tumor cohorts - Melanoma, HCC and RCC.
  Interventions: Drug: HBM4003

INTERVENTIONS:
Drug: HBM4003 — Intravenous (IV) administration

SUMMARY:
This is a study to evaluate the safety and tolerability of the study drug HBM4003, and to determine the maximum tolerated dose and/or recommended Phase 2 study dose of HBM4003. The study will also look at the anti-tumor activity of HBM4003.The study consists of 2 parts. In Part 1, patients are enrolled into different cohort doses in order to identify the appropriate recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD). In Part 2, participants with metastatic/unresectable melanoma will receive the MTD and/or RP2D established in Part 1 of the study. In Part 1 and Part 2, participants will be administered treatment either once per week or once every 3 weeks.

NOTE: Participants are no longer being recruited to this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form and willingness to comply with study requirements.
* Part 1 (Dose-escalation): Adult subject ≤ 75 years old with confirmed advanced solid tumors that have progressed after treatment with standard therapies, or for which no effective standard therapy is available, or the subject refuses or has a contraindication to standard therapy.
* Part 2 (Dose-expansion)

  * Adult subjects 18 years and above.

Melanoma Cohort:

1. Histologically confirmed metastatic or unresectable melanoma that progressed during or after treatment with a PD-1 inhibitor (excluding bi-specific antibody) with CTLA-4 blocking function.
2. Must have received at least one BRAF inhibitor with/without a MEK inhibitor if positive with BRAF V600-activating mutation.

HCC Cohort:

1. Histologically confirmed metastatic or unresectable hepatocellular carcinoma;
2. Child-Pugh Score of 6 points or less (A5-A6);
3. Patient with HBV infection will be allowed if he/she is receiving appropriate antiviral therapy for hepatitis B virus (HBV) according to institutional standard of care and HBV DNA level is < 2000 UI/mL;
4. Patient with HCV infection will be allowed if he/she is receiving appropriate antiviral therapy for hepatitis C virus (HCV) according to institutional standard of care and HCV antibody returns to negative;
5. Have received at least one anti-VEGF treatment (either anti-VEGFR TKI or anti-VEGF monoclonal antibody) and/or anti-PD-(L)1 treatment.

RCC Cohort:

1. Histologically confirmed metastatic or unresectable renal cell cancer (including both clear cell and non-clear histology);
2. Subjects with clear cell RCC must have failed at least 1 anti-VEGFR TKI treatment and/or anti-PD(L)1 treatment;
3. For subjects with non-clear cell RCC (e.g. PRCC), treatment naive is permitted.

   * Must have at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
   * Willing to undergo tumor biopsy unless determined medically unsafe or not feasible.
   * For subjects whose last treatment was immunotherapy, must have disease progression confirmed at least 4 weeks after the initial radiographic evidence of progression;
   * Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
   * Adequate organ and bone marrow function.
   * Females of childbearing potential may participate provided they agree to practice abstinence; and, if heterosexually active, agree to use at least 2 highly effective contraceptive methods throughout the study and for 3 months following the last dose of HBM4003; and have a negative serum pregnancy test.
   * Females of non-childbearing potential must be post-menopausal or have been surgically sterilized.
   * Male subjects with a female partner of childbearing potential must agree to practice abstinence or to use a physician-approved contraceptive method throughout the study and for 3 months following the last dose of study drug.
   * Life expectancy of ≥12 weeks.

Exclusion Criteria:

Part 1 and Part 2

* History of severe or not under well controlled allergic diseases, history of severe drug allergy, or are known to be allergic to macromolecular protein preparations or any component of the study drug.
* Receipt of anticancer medications or investigational drugs within the following intervals before the first administration of the study drug:

  1. CTLA-4 antibody any time prior to study drug administration;
  2. Any PD-1 or PD-L1 or Programmed cell death protein ligand 2 (PDL2)-directed antibody within 8 weeks of study drug administration;
  3. Any cancer vaccines within 3 months prior to first dose of study drug;
  4. Live vaccine within 4 weeks prior to first dose of study drug;
  5. Any other anticancer therapy within 2 weeks prior to first dose of study drug.
* Not yet recovered from surgery within 28 days prior to first dose of HBM4003 or (immune-related) toxicity related with previous treatment.
* Concomitant medication or treatments:

  1. Any concurrent chemotherapy, radiotherapy, immunotherapy, or biological therapy for cancer treatment. Concurrent use of hormones on a stable dose for non-cancer related conditions is acceptable. Androgen deprivation therapy (ADT) for advanced prostate cancers is acceptable. Local treatment of isolated non-target lesions for palliative intent is acceptable;
  2. Any traditional anti-tumor herbal medications;
  3. Receipt of red blood cells or platelets infusion, granulocyte colony stimulating factor (G-CSF) or granulocyte monocyte colony stimulating factor (GM-CSF) within 1 week of the first dose of HBM4003.
  4. Corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 2 weeks of study drug administration; Nasal spray, inhalation, topical corticosteroids or physiological doses of systemic corticosteroids are not included.
* Have other diseases that may affect the effectiveness and safety of the study drug, such as:

  1. Known brain metastases or other central nervous system metastases that is either symptomatic or untreated, that requires concurrent treatment;
  2. Active infection requiring treatment with antibiotics within 14 days prior to first dose of HBM4003;
  3. Known history of infection with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), human T lymphotropic virus 1, hepatitis B virus, or active hepatitis C virus;
  4. Suspected autoimmune disease, including but not limited to inflammatory bowel disease, autoimmune hepatitis, Guillain-Barre syndrome.
  5. Known primary immunodeficiency;
  6. Clinically significant gastrointestinal disorders (e.g. diarrhea with significant clinical meaning), active gastrointestinal bleeding, or a history of gastrointestinal perforation, acute diverticulitis, intra-abdominal abscess or gastrointestinal obstruction;
  7. Have received allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or have received autologous hematopoietic stem cell transplantation within 3 months prior to the first dose of study drug.
  8. Subjects with medically confirmed autoimmune coeliac disease are to be excluded. Patients with so-called gluten intolerance or other conditions labelled "coeliac disease" which are not autoimmune in nature and which are well controlled by diet should be medically confirmed as non-autoimmune "coeliac disease" and can be considered for study.
* Subjects with major cardiovascular disease.
* History of other uncured malignant diseases, except for non-melanoma skin cancer in situ, superficial bladder cancer, cervical cancer in situ that has been curatively resected, and localized prostate cancer managed by active surveillance.
* Pregnant or breastfeeding women.
* Have experienced immune-related GI adverse events on any prior immunotherapy or toxicity that led to permanent discontinuation of prior immunotherapy.
* Severe cirrhosis, hepatic atrophy, portal hypertension.
* Main portal vein thrombosis present on imaging.
* Any prior or current clinically significant ascites (moderate to massive with significantly abnormal liver function).
* Any history of hepatic encephalopathy within 12 months prior to randomization or require medications to prevent or control encephalopathy.
* Subjects weighting < 30 kg.
* Active or prior documented GI bleeding (e.g. esophageal varices or ulcer bleeding) within 12 months.

Additional criterial for HCC cohort:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Prior liver transplantation.
* HBV and HCV co-infection, HBV and HEV co-infection, HBV and HDV co-infection.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Part 1: Proportion of subjects with Dose-Limiting Toxicity (DLT) | From Day 1 until disease progression or Day 28, whichever comes first
  Number of subjects who experience DLT events during 28 days (if on QW dosing schedule) or 21 days (if on Q3W dosing schedule)
Part 2: Objective Response Rate (ORR) | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Proportion of subjects with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1

SECONDARY OUTCOMES:
Part 1: Objective Response Rate | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Proportion of subjects with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1
Part 1: Duration of response | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Time interval from first occurrence of a documented objective response to the time of disease progression, as determined by the Investigator using RECIST 1.1 or death from any cause, whichever comes first.
Part 1: Disease control rate | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Proportion of subjects with a best overall response of complete response (CR), partial response (PR) or stable disease (SD).
Part 1: Duration of disease control | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Time from data of start of treatment to the date of disease progression or death for subjects who had CR or PR or SD during treatment.
Part 1: Tumor shrinkage (The percentage of patients with tumor shrinkage) | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Greatest tumor shrinkage achieved at any follow-up assessment. Measured by radiological (computed tomography [CT]/Magnetic Resonance Imaging [MRI]) scanning until documented radiographic disease progression according to RECIST 1.1, or loss of clinical benefit after disease progression according to RECIST 1.1
Part 1: Cmax (Maximum serum concentration) | Up to 80 days after end of treatment
Part 1: Tmax (Time to reach maximum serum concentration) | Up to 80 days after end of treatment
  Plasma
Part 1: AUC0-inf (Area under the serum concentration versus time curve from time zero to infinity | Up to 80 days after end of treatment
Part 1: Vss (Volume of distribution at steady state) | Up to 80 days after end of treatment
  Amount of drug in the body divided by plasma concentration
Part 1: AUC0-tau (Area under the serum concentration versus time curve from time zero to the dosing interval tau | Up to 80 days after end of treatment
Part 1: t1/2 (Terminal half-life) | Up to 80 days after end of treatment
Part 1: Clearance (CL) | Up to 80 days after end of treatment
Part 1: Cmin (Minimum serum concentration) | Up to 80 days after end of treatment
  Minimum blood plasma concentration reached by drug prior to administration of second dose
Part 1: Rac(Cmax) | Up to 80 days after end of treatment
  Accumulation ratio calculated from Cmax,ss (maximum (peak) steady state plasma drug concentration during a dosage interval) and Cmax after single dosing
Part 1: Rac(AUC0-tau) | Up to 80 days after end of treatment
  Accumulation ratio calculated from AUCτ,ss and AUC after single dosing
Part 2: Disease control rate | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Proportion of subjects with a best overall response of complete response (CR), partial response (PR) or stable disease (SD).
Part 2: Duration of objective response | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Time interval from first occurrence of a documented objective response to the time of disease progression, as determined by the Investigator using RECIST 1.1 and iRECIST, or mRECIST for hepatocellular carcinoma (HCC)
Part 2: Objective Response Rate | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Proportion of subjects with best overall response of complete response (CR) or partial response (PR) per Response Criteria for Use in Trials Testing Immunotherapeutics (iRECIST), or modified RECIST (mRECIST) for HCC
Part 2: Duration of disease control | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Time from data of start of treatment to the date of disease progression or death for subjects who had CR or PR or SD during treatment.
Part 2: Tumor shrinkage (The percentage of patients with tumor shrinkage) | Up to day 206 or until disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefit, death or termination of study, whichever comes first.
  Greatest tumor shrinkage achieved at any follow-up assessment. Measured by radiological (computed tomography [CT]/Magnetic Resonance Imaging [MRI]) scanning until documented radiographic disease progression according to RECIST 1.1, or loss of clinical benefit after disease progression according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (17):
- Australia (4):
  - St. George Private Hospital, 1 South Street, Kogarah, New South Wales
  - Macquarie University, 2 Technology Place, Macquarie, New South Wales
  - Monash Health, Monash Medical Centre, 246 Clayton Road, Clayton, Victoria
  - The Alfred Hospital, Commercial Road, Melbourne, Victoria
- China (12):
  - Union Hospital affiliated to Tongji Medical College of HUST, Oncology Department, No. 1277 Jiefang Dadao, Wuhan, Hubei
  - Yantai Yuhuangding Hospital, Urology Department, 8th Floor, No. 20 Donglu Road, Zhifu District, Yantai, Shandong
  - The Second People's Hospital of Yibin, Oncology Department, No. 268 South Bank Nanguang Road, Xuzhou District, Yibin, Sichuan
  - Zhejiang Cancer Hospital, Department of Head and Neck Medicine for Rare Diseases, No. 1, Banshan Road, Gongshu District, Hangzhou, Zhejiang
  - Zhenjiang Cancer Hospital, Department of Interventional Therapy, No. 1, Banshan Road, Gongshu District, Hangzhou, Zhejiang
  - Peking University First Hospital, Chemotherapy Department, No. 15 cheniandian Hutong, Annei Street, Dongcheng District, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Oncology Department, No. 17 Panjiayuan Nanli, Chaoyang District, Beijing
  - Hunan Cancer Hospital, Intervention Division, 83 Tongzipo Road, Yuelu District, Changsha
  - Hunan Cancer Hospital, Urology Department, 83 Tongzipo Road, Yuelu District, Changsha
  - Tianjin Medical University Cancer Institute and Hospital, Biotherapeutic Department, 17 / F, Block C, West Huan-Hu Rd., Ti Yuan Bei, Hexi District, Tianjin
  - Xuzhou Central Hospital, Oncology Department, No. 199 Jiefang South Road, Quanshan District, Xuzhou
  - Henan Cancer Hospital, Oncology Department, No. 127 Dongming Road, Jinshui District, Zhengzhou
- Queen Mary Hospital, Department of Medicine, 102 Pok Fu Lam Road, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data generated by this study will be considered confidential by the Investigator, except to the extent that it is included in a publication. The general strategy regarding publication of the study will be mutually agreed upon by the Investigator and Sponsor. The Sponsor reserves the right to manage the publication of all study results. The Investigator agrees that oral and written communication to third parties of any procedures or results from the study is subject to prior written consent of the Sponsor. Presentation material and/or manuscript(s) for publication will be reviewed by the Sponsor prior to submission for publication. Alterations in the material will only be made in agreement between the Investigator and the Sponsor.

REFERENCES:
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts